CLINICAL TRIAL: NCT00553046
Title: Italian Multicenter Survey on the Last 3 Months of Life in Patients Ventilated at Home
Brief Title: Last 3 Months of Life in Home Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Michele Vitacca, Principal Investigator, Fondazione Salvatore Maugeri
Other Study IDs: N°159
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2007-10

CONDITIONS: Respiratory Failure
Keywords: ethics; COPD; end of life; mechanical ventilation; CRF home ventilated patients
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Death | interventions — Zarit Caregiver Burden Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- family burden: chronich respiratory failure home ventilated patients
  Interventions: Other: survey administration

INTERVENTIONS:
Other: survey administration — application of a family survey on last 3 months of life for their relatives under HMV
  Other Names: caregiver burden

SUMMARY:
To verify with a specific questionnaire, the families' perceived quality of end-of-life care and of dying in the last 3 months of life of 168 patients (Chronic Obstructive Pulmonary Disease-Amyotrophic Lateral Sclerosis (ALS)-Restrictive disorders-Neuromuscular disease- others) with chronic respiratory failure needing domiciliary mechanical ventilation (MV).

DETAILED DESCRIPTION:
Participants: 168 patients' relatives presenting five categories of diseases (Chronic Obstructive Pulmonary Disease-Amyothrophic Lateral Sclerosis (ALS)-Restrictive disorders-Neuromuscular disease- others) answered to questionnaire.

Interventions: none Measurements and Main Results: 35 questions grouped in 6 specific domains (Control of pain and symptoms (domain 1-D1), awareness of disease (D2), family burden (D3), the process of dying (D4), medical troubles including hospitalizations (D5) and technical problems linked to MV(D6) were asked after the patient's death to a family member by means of a face to face interview. Answers to the binary 35-item questionnaire were distributed into just two clusters per each domain.

ELIGIBILITY:
Inclusion criteria:

All patients mechanically ventilated at home who died

Exclusion criteria:

patients with cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Home MV patients in the last 3 months of life
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
level of family burden | 3 months after patient's death

SECONDARY OUTCOMES:
influence of diagnosis and modality of ventilation | 3 months after patient's death

CONTACTS AND LOCATIONS:
Overall Officials: michele vitacca, MD, Principal Investigator — Fondazione S. Maugeri IRCCS
Locations (1):
- FSM Respiratory Unit, Lumezzane, BS, Italy

REFERENCES:
- [Background] Singer PA, Martin DK, Kelner M. Quality end-of-life care: patients' perspectives. JAMA. 1999 Jan 13;281(2):163-8. doi: 10.1001/jama.281.2.163. PMID 9917120
- [Result] Vitacca M, Comini L & Barbano L. Home mechanical ventilation difficulties in the last 3 months of life as reported by caregivers. J Med Pers 11:30-36, 2013. DOI 10.1007/s12682-012-0128-8